CLINICAL TRIAL: NCT05485766
Title: Neoadjuvant and Adjuvant Olaparib Plus Pembrolizumab Following Platinum Based Chemotherapy Plus Pembrolizumab for Germline BRCA Mutated Triple Negative Breast Cancer (WJOG14020B/OPERETTA)
Brief Title: Novel Neoadjuvant and Adjuvant Strategy for Germline BRCA 1/2 Mutated Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Okayama University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yuko Takahashi, Assistant professor, Endocrinological Center, Okayama University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUMK59829
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Triple Negative Breast Neoplasms; Triple Negative Breast Cancer; Breast Neoplasms; Breast Cancer; BRCA1 Mutation; BRCA2 Mutation; BRCA Mutation; BRCA-Associated Breast Carcinoma
Keywords: BRCA1 protein; BRCA2 protein
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — pembrolizumab; Paclitaxel; Carboplatin; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab+ Paclitaxel + Carboplatin Followed by Pembrolizumab + Olaparib (Experimental): 1. Neoadjuvant phase; Treatment 1: Pembrolizumab+ Paclitaxel + Carboplatin (Cycles 1-4) Treatment 2: Pembrolizumab + Olaparib (Cycles 1-4)
  2. Definitive Surgery
  3. Adjuvant phase; Pembrolizumab + Olaparib (1-9 cycles)
  Note: each cycle = 3 weeks (Neoadjuvant Treatment 1 and 2, and Adjuvant Treatment)
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Olaparib; Procedure: Definitive Surgery

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg fixed dose, IV, every 3 weeks (Q3W), on Days 1 of Cycles 1-4
  Other Names: Keytruda; MK-3475
Drug: Paclitaxel — 80 mg/m2, IV, weekly, on Days 1, 8, 15 of Cycles 1-4
Drug: Carboplatin — Area under the curve (AUC 1.5), intravenously (IV), weekly, on Days 1, 8, 15 of Cycles 1-4
Drug: Olaparib — 300 mg BID (twice daily) orally
  Other Names: Lynparza
Procedure: Definitive Surgery — Each subject will undergo definitive surgery 3-6 weeks after conclusion of the last cycle of the neoadjuvant treatment.

SUMMARY:
This is a Phase II, single-arm, open label study to evaluate Olaparib plus Pembrolizumab following platinum-based chemotherapy plus Pembrolizumab as neoadjuvant therapy for germline BRCA (gBRCA) 1/2 mutated triple negative breast cancer (TNBC).

Pembrolizumab in combination with weekly paclitaxel and carboplatin (treatment 1) is followed by Pembrolizumab in combination with Olaparib (treatment 2) in neoadjuvant setting and Pembrolizumab in combination with Olaparib in adjuvant setting will be studied

ELIGIBILITY:
Inclusion Criteria:

* Male/female subjects who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of invasive breast cancer
* Have histologically confirmed TNBC, as defined by the most recent ASCO/CAP guidelines.
* Confirmed germline BRCA 1/2 mutated.
* Have previously untreated locally advanced non-metastatic (M0) TNBC defined as the following combined primary tumor (T) and regional lymph node (N) staging per AJCC for breast cancer staging criteria version 7 as assessed by the investigator based on radiological and/or clinical assessment:

  1. T1c, N1-N2
  2. T2, N0-N2
  3. T3, N0-N2
  4. T4a-d, N0-N2
* It has been confirmed that there is no distant metastasis to each organ by the following tests. Chest: Contrast CT or FDG-PET/CT Abdominal: Contract CT* or FDG-PET/CT Bone: Bone scintigraphy or FDG-PET/CT Brain: In the case of no central nervous system symptoms, examination for brain metastasis is not required.
* The subject (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Have adequate organ function as defined in the protocol. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

* Subjects who has a positive urine pregnancy test within 72 hours prior to registration
* Has diagnosed as inflammatory breast cancer.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor .
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and investigational drugs used in this study and/or any of their excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (non-infectious) pneumonitis/interstitial lung disease .
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HbsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children.
* Has had an allogenic tissue/solid organ transplant.
* Has received pre-treatment with Olaparib or other PARP inhibitors.
* Has significant cardiovascular disease
* Has a resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions.
* Subject has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Subject received colony-stimulating factors within 28 days prior to the first dose of study intervention.
* Subject is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* Is either unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption.
* Is, in the judgement of the investigator, unlikely to comply with the study procedures, restrictions, and requirements of the study.
* Is currently receiving either strong or moderate inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study.
* Is currently receiving either strong or moderate inducers of CYP3A4 that cannot be discontinued for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate (ypT0/TisypN0) | From 27 weeks up to 30 weeks
  Pathological complete response rate (ypT0/TisypN0) is defined as the proportion of subjects without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by AJCC staging criteria (7th edition) assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Residual Cancer Burden 0/1 | From 27 weeks up to 30 weeks
  Residual Cancer Burden (RCB) 0/1 rate is defined as the proportion of subjects on evaluation from routine pathologic sections of the primary breast tumor and the regional lymph nodes after the completion of neoadjuvant therapy assessed by the local pathologist at the time of definitive surgery. Six variables are included in a calculation formula. The calculated RCB index value can also be categorized as one of four RCB classes (0 - 3). The calculation formula and detailed description can be found at a dedicated Web site: http://www.mdanderson.org/breastcancer_RCB.
Pathological Complete Response (pCR) Rate (ypT0/is) | From 27 weeks up to 30 weeks
  Pathological complete response rate (ypT0/is) is defined as the proportion of subjects without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen regardless of regional lymph nodes status following completion of neoadjuvant systemic therapy by AJCC staging criteria (7th edition) assessed by the local pathologist at the time of definitive surgery.
Pathological Complete Response (pCR) Rate (ypT0/Tis ypN0) | From 27 weeks Up to 30 weeks
  Pathological complete response rate (ypT0/TisypN0) is defined as the proportion of subjects without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by AJCC staging criteria (7th edition) assessed by the local pathologist at the time of definitive surgery.
Three-Year Overall Survival (3-year OS) | Up to 3 years
  The Proportion of Three Year-Overall Survival (3y-OS) is defined as the proportion of survival subjects without death due to any cause at 3 years from registration. Subjects without documented death at the time of the analysis will be censored at the date of the last follow-up.
Three-Year Distant Metastatic Free Survival (3-year DMFS) | Up to 3 years
  The Proportion of Three-Year Distant Metastatic Free Survival (3y-DMFS) is defined as the proportion of survival subjects without distant metastatic disease at 3 years from registration. Subjects without documented distant metastatic disease at the time of the analysis will be censored at the date of the last follow-up.
Three-Year Disease Free Survival (3-year DFS) | Up to 3 years
  The Proportion of Three-Year Disease Free Survival (3y-DFS) is defined as the proportion of survival subjects without metastatic disease and secondary malignancy at 3 years from registration. Subjects without documented metastatic disease and secondary malignancy at the time of the analysis will be censored at the date of the last follow-up.
AEs/SAEs and treatment discontinuation due to AEs/SAEs | Up to 3 years
  Safety measurements are the incidence of, causality of, and outcome of AEs/SAEs; and changes in vital sign measurements and laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Takahashi, MD., PhD., Principal Investigator — Assistant Professor, Endocrinological Center, Okayama University Hospital
Locations (3):
- Japan (3):
  - Gifu University Hospital, Gifu, Gifu
  - Okayama University Hospital, Okayama
  - St. Luke's International Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No